CLINICAL TRIAL: NCT05786846
Title: Serum Thyroid Function After Iodinated Contrast Administration in Chinese Euthyroid Adults: a Prospective Observational Study.
Brief Title: Serum Thyroid Function After Iodinated Contrast Administration
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSEC-KY-KS-2022-002
Record Dates: First submitted 2023-02-16; First posted 2023-03-28 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-02

CONDITIONS: Thyroid Dysfunction
MeSH Terms: interventions — Diatrizoate Meglumine; iopromide; Iohexol; ioversol; Iopamidol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Iodinated contrast agents — Patients who use iodinated contrast agents clinically
  Other Names: Meglumine diatrizoate; Iopromide; Iohexol; Ioversol; Iopamidol

SUMMARY:
This study investigated the changes in serum thyroid function and urinary iodine levels before and after the use of iodinated contrast to analyze the prevalence of thyroid dysfunction in the Chinese euthyroid adults after using iodinated contrast.

DETAILED DESCRIPTION:
This study aims to monitor the thyroid function, urinary iodine level, and other indicators of patients after using iodine contrast agents, in order to analyze the prevalence of thyroid dysfunction after using iodine containing contrast agents, and investigate the impact of different iodine contrast agents on thyroid function, in order to provide evidence for the use of iodine contrast agents in clinical practice and the risk prevention of subsequent thyroid diseases.

ELIGIBILITY:
Inclusion Criteria:

* patients who use iodinated contrast agent

Exclusion Criteria:

* patients with the following diseases: malignant tumor, critical illness (admitted to ICU), mental disease, hypothalamus-pituitary disease.
* administration of anti-thyroid drugs (methimazole, propylthiouracil), levothyroxine, compound iodine solution, amiodarone, immunostaining point inhibitor, tyrosine kinase inhibitor, interferon, interleukin-6, lithium, glucocorticoids β Receptor blockers, dopamine, dobutamine, bromocriptine, octreotide, phenobarbital, phenytoin sodium, rifampicin, and carbamazepine within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are identified of having undergone a radiological examination use of an iodinated contrast agent in Sun Yat-sen Memorial Hospital of Sun Yat-sen University
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of thyroid dysfunction after administration of iodine contrast agent. | up to 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Li Yan, Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No